CLINICAL TRIAL: NCT01463475
Title: University of Wisconsin hMSC Cell Bank: Bone Marrow Donor Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: H-2010-0104; HHSN268201000010C (Other Grant/Funding Number: NATIONAL HEART, LUNG, AND BLOOD INSTITUTE)
Record Dates: First submitted 2011-09-30; First posted 2011-11-02 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Graft Versus Host Disease (GVHD); Acute Myocardial Infarction (AMI)
Keywords: MSC; Allogeneic; Bone marrow cells; Healthy subject donors; Collection of MSC from bone marrow aspirate; Bronchiolitis obliterans syndrome (BOS)
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bone Marrow Aspirate (Other): A qualified enrolled donor will have an aspirate bone marrow draw.
  Interventions: Procedure: Bone marrow aspirate

INTERVENTIONS:
Procedure: Bone marrow aspirate — A single bone marrow aspirate procedure is planned.
  Other Names: bone marrow-derived MSC

SUMMARY:
The objective of this protocol is to use established standard criteria and methods for the collection of hMSC (human mesenchymal stromal cells) from healthy bone marrow donors. The hMSC collected from the donors will use to develop well-defined and reproducible cell banks. Standard manufacturing procedures and quality control testing methods will be used to characterize and evaluate the final cell product. After the cell banks are created, these cell products will be used in future translational or clinical research.

DETAILED DESCRIPTION:
Cell banks will be manufactured and cellular products used for future translational or clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 35 years
* Willingness to provide written informed consent

Exclusion Criteria:

* Presence of risk factors for or clinical evidence of Human immunodeficiency virus (type 1 and 2), Hepatitis B, Hepatitis C, Human T-lymphotrophic virus (type I and II), Human transmissible spongiform encephalopathy (including Creutzfeldt-Jakob disease) treponema pallidum,
* Presence of communicable disease risk associated with xenotransplantation.
* Test positive for Human immunodeficiency virus (type 1 and 2), Hepatitis B, Hepatitis C, Human T-lymphotrophic virus (type I and II), cytomegalovirus (CVM), West Nile Virus, treponema pallidum.
* Use of investigational drug within 30 days or 5 half lives which ever is longer. Use of investigational implanted device.
* History of malignancy.
* Pregnancy
* In the opinion of the hematologist or the investigator, a condition that compromises the ability of the donor to safely provide BM donation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Culture and expand mesenchymal stromal cells (MSC) | Day 1- cells are counted within 24 hours of bone marrow aspirate collection
  Cell viability, proliferation profile, and expression characteristics will be evaluated.

SECONDARY OUTCOMES:
Characterization profile of MSC during and after expansion will be assessed | Examine the cell surface marker profile of MSC using standard flow cytometry
  Cell surface expression profile will be obtained using Flow Cytometry. Additional characterization includes cell differentiation profile.

CONTACTS AND LOCATIONS:
Overall Officials: Peiman Hematti, MD, Principal Investigator — University of Wisconsin, Madison; John M Centanni, MS, Study Director — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States